CLINICAL TRIAL: NCT06393868
Title: Reducing Gastrointestinal Bleeding With Proton Pump Inhibitor Therapy in Acute Venous Thromboembolism: Pilot Randomized Study (RADIANT Study)
Brief Title: Reducing Gastrointestinal Bleeding With Proton Pump Inhibitor Therapy in Acute Venous Thromboembolism
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RADIANT-001
Record Dates: First submitted 2024-03-19; First posted 2024-05-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Venous Thromboembolism; Gastro Intestinal Bleeding; Blood Clot
Keywords: Omeprazole; VTE; GI Bleeding
MeSH Terms: conditions — Venous Thromboembolism; Gastrointestinal Hemorrhage; Thrombosis | interventions — Omeprazole; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily dose of omeprazole 20 mg (Experimental): Participants randomized to the experimental arm will take one omeprazole 20 mg tablet by mouth every day for the duration of their participation in the study.
  Interventions: Drug: Omeprazole 20 mg Oral Tablet
- Daily dose of placebo (Placebo Comparator): Participants randomized to the control arm will take one placebo tablet by mouth every day for the duration of their participation in the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omeprazole 20 mg Oral Tablet — Omeprazole once daily for 90 days
  Other Names: Omeprazole
  Arms: Daily dose of omeprazole 20 mg
Other: Placebo — Placebo once daily for 90 days
  Arms: Daily dose of placebo

SUMMARY:
The investigators are studying whether treatment with a proton pump inhibitor called omeprazole reduces gastrointestinal bleeding in older adults taking blood thinners for a blood clot (venous thromboembolism). The purpose of this study, a pilot study or a feasibility study, is to test the study plan and determine whether enough participants will join a larger study and accept the study procedures.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) refers to blood clots that form in the veins of the body, including the arms or legs (deep vein thrombosis [DVT]), abdomen (portal vein thrombosis), or lungs (pulmonary embolism [PE]). These blood clots are treated with medication to reduce blood clotting called anticoagulants. The main complication of anticoagulants is bleeding, the majority of which comes from the stomach or intestines (gastrointestinal tract). Anticoagulants do not cause bleeding, but they may make bleeding worse. Uncommonly, serious gastrointestinal (GI) bleeding can happen leading to hospitalization and even death. The chance of bleeding is highest in the first few months after starting anticoagulants.

Proton pump inhibitors (PPIs) are medications that lower the acid content of the stomach. The medication in this study, a type of proton pump inhibitor called omeprazole, is approved in Canada for treating stomach ulcers, heartburn, and a stomach infection called Helicobacter pylori. The use of omeprazole in this study is considered investigational. This means that Health Canada has not approved the use of omeprazole as a treatment for preventing gastrointestinal bleeding in patients taking anticoagulants. Some studies suggest that they may reduce gastrointestinal bleeding for people taking anticoagulants.

The investigators are studying whether treatment with a proton pump inhibitor called omeprazole reduces gastrointestinal bleeding in older adults taking anticoagulants for venous thromboembolism.

The investigators plan to do a large, randomized trial which is the best way to test the effect of a treatment. To do this, some of the participants in this study will get omeprazole and others will get a placebo (a substance that looks like the study omeprazole but does not have any active or medicinal ingredients). The placebo in this study is not intended to have any effect on bleeding. A placebo is used to make the results of the study more reliable.

Primary Objective To assess the feasibility of a full-scale double-blind placebo-controlled randomized trial to determine whether omeprazole reduces the risk of upper GI bleeding in older adults receiving anticoagulation for acute VTE compared to placebo.

Secondary Objectives:

1. To measure additional feasibility outcomes
2. To measure informative outcomes
3. To measure key clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 65 years or older at the time of enrolment. Enrolment is limited to older adults as age is an important non-modifiable risk factor for bleeding. This will ensure the study population includes participants who may be more likely to benefit from omeprazole (compared to those with no risk factors) because all participants will have at least 1 risk factor for bleeding.
2. Newly diagnosed VTE which includes VTE at any site such as (but not limited to) DVT of upper or lower limbs, PE, cerebral vein thrombosis, portal vein thrombosis, other splanchnic vein thrombosis.
3. Planned for 3 months (90 days) or more of therapeutic anticoagulation with any anticoagulant.
4. Patient or delegate is able and willing to comply with follow-up examinations contained within the consent form.

Exclusion Criteria:

1. Therapeutic anticoagulation therapy for more than 7 days
2. Currently prescribed PPI for regular daily use (patients receiving H2 receptor antagonists will not be excluded),
3. Previous upper GI bleeding,
4. Need for dual antiplatelet therapy,
5. Contraindications to omeprazole (hypersensitivity to omeprazole, or other substituted benzimidazole PPIs, concomitant use with products that contain rilpivirine, significant drug interactions, up to the discretion of the site investigator),
6. Life expectancy is less than 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Study feasibility at participating centres | 24 months
  The mean number of participants recruited per site per month

SECONDARY OUTCOMES:
Eligibility Rate | 24 months
  Proportion of screened patients who are eligible
Consent Rate | 24 months
  Proportion of eligible patients who provide consent
Retention Rate | 27 months
  Proportion of participants who completed all study procedures
Adherence Rate | 27 months
  adherence to study drug measured by pill count or assessing the patient diary at the end of follow-up

OTHER OUTCOMES:
Risk Factors | 24 months
  The proportion of participants with the following risk factors for bleeding at baseline: decreased kidney function (defined as estimated glomerular filtration rate [eGFR] <60 mL/min/1.73 m2), active cancer, concurrent antiplatelet and/or NSAID therapy, chronic liver disease, chronic anemia.
Patients already prescribed proton pump inhibitor | 24 months
  The proportion of screened patients already receiving prescribed proton pump inhibitor therapy
Reasons for Declining Participation | 24 months
  Patients are not required to provide a reason for declining to participate. However, for those patients who are willing to share, reasons for declining participation will be reviewed
New PPI prescription | 27 months
  The proportion of participants with new prescription for proton pump inhibitor during the study
Recurrent VTE | 27 months
  The proportion of patients that have a recurrent venous thromboembolism during the study
Mortality | 27 months
  The proportion of patients who die from gastrointestinal bleeding, and all-cause mortality during the study
Serious Adverse Events | 27 months
  The proportion of patients who have a serious adverse event during the study
Change in health-related quality of life | 27 months
  Change in health-related quality of life as measured by the EuroQol EQ-5D-5L Quality of Life questionnaire at 90 days compared to baseline. This questionnaire includes the patient's thoughts about their health, including mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. The lowest possible score is 5 and the highest is 25. A lower score represents a worse quality of life. The questionnaire also includes a Visible Analog Scale where patients are asked to picture a vertical line that is numbered from 0 to 100. 100 at the top of the line means the best health the patient can imagine and 0 at the bottom of the line means the worst health the patient can imagine. Patients are asked to provide a number that best represents their health at the time of completing the questionnaire.
Change in functional status | 27 months
  Change in functional status as measured by the Standard Assessment of Global Activities in the Elderly (SAGE) scale at 90 days compared to baseline. The SAGE questionnaire measures what patients are doing in their community and their homes. Patients are asked to indicate the level of difficulty they have with each of the questions in the past month with a response of no difficulty, mild, moderate, or severe difficulty. Mild = minimal/occasional difficulty that does not affect the ability to perform the activity or task; Moderate = some/regular difficulty that does affect the ability to perform the task, although they may still be able to perform the task; Severe = extreme/constant difficulty performing the task or the task is not completed and/or is completed by someone else because of its difficulty.
Clinically Relevant Upper Gastrointestinal Bleeding Events | 27 months
  Adjudicated clinically relevant upper gastrointestinal bleeding (major upper gastrointestinal bleeding plus clinically relevant non-major [CRNM] upper GI bleeding, adapted from International Society on Thrombosis and Haemostasis (ISTH) criteria for major bleeding and CRNM bleeding).
Rate of endoscopically confirmed upper gastrointestinal bleeding | 27 months
  Proportion of patients who have upper gastrointestinal bleeding as confirmed by endoscope at 30, 60, and 90 days post randomization
Rate of lower gastrointestinal bleeding | 27 months
  Proportion of patients who have lower gastrointestinal bleeding at 30, 60, and 90 days post randomization
All major gastrointestinal bleeding | 27 months
  Proportion of patients who have confirmed major gastrointestinal bleeding by adjudication at 30, 60, and 90 days post randomization
All clinically relevant non-major gastrointestinal bleeding | 27 months
  Proportion of patients who have confirmed clinically relevant non-major gastrointestinal bleeding by adjudication at 30, 60. 90 days
All major bleeding | 27 months
  Proportion of patients who have confirmed major bleeding by adjudication, including major GI bleeding) at 30, 60, 90 days post randomization
All clinically relevant non-major bleeding | 27 months
  Proportion of patients who have confirmed clinically relevant non-major bleeding (including CRNM GI bleeding) at 30, 60, and 90 days post randomization
Hospitalization for gastrointestinal bleeding | 27 months
  Proportion of patients hospitalized for gastrointestinal bleeding at 30, 60. and 90 days post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Siegal, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (7):
- Canada (7):
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System - St. Catharines Site, St. Catharines, Ontario
  - University Health Network - Toronto General, Toronto, Ontario
  - CIUSSS de l'Est-de- l'Île-de-Montréal, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU de Québec-Université Laval; Hôpital Saint-François d'Assise, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
CONVERGE trials will be conducted within specific research domains under a core protocol outlining shared elements, including broad inclusion criteria, a minimum set of core outcomes, event adjudication, and data sharing to the CONVERGE shared data repository. Patients meeting domain-specific inclusion criteria can be enrolled in individual trials based on pre-defined additional characteristics. RADIANT will be the first trial conducted within the Acute VTE Treatment Domain.
Supporting Information: Study Protocol
Time Frame: Starting after study completion
Access Criteria: Select members of the International Network of VENous Thromboembolism Clinical Research Networks (INVENT) participating in CONVERGE trials will enter into an agreement to enhance data-sharing and meta-analysis across trials. Access will be restricted by strict authentication processes and data will be maintained on secure servers.

REFERENCES:
- [Background] Wendelboe AM, McCumber M, Hylek EM, Buller H, Weitz JI, Raskob G; ISTH Steering Committee for World Thrombosis Day. Global public awareness of venous thromboembolism. J Thromb Haemost. 2015 Aug;13(8):1365-71. doi: 10.1111/jth.13031. Epub 2015 Jul 14. PMID 26084415
- [Background] Delluc A, Tromeur C, Le Ven F, Gouillou M, Paleiron N, Bressollette L, Nonent M, Salaun PY, Lacut K, Leroyer C, Le Gal G, Couturaud F, Mottier D; EPIGETBO study group. Current incidence of venous thromboembolism and comparison with 1998: a community-based study in Western France. Thromb Haemost. 2016 Oct 28;116(5):967-974. doi: 10.1160/TH16-03-0205. Epub 2016 Jul 28. PMID 27465905
- [Background] Heit JA. Epidemiology of venous thromboembolism. Nat Rev Cardiol. 2015 Aug;12(8):464-74. doi: 10.1038/nrcardio.2015.83. Epub 2015 Jun 16. PMID 26076949
- [Background] Heit JA, Spencer FA, White RH. The epidemiology of venous thromboembolism. J Thromb Thrombolysis. 2016 Jan;41(1):3-14. doi: 10.1007/s11239-015-1311-6. PMID 26780736
- [Background] Ferrazzini E, Mean M, Stalder O, Limacher A, Rodondi N, Aujesky D. Incidence and clinical impact of bleeding events in older patients with acute venous thromboembolism. Blood Adv. 2023 Jan 24;7(2):205-213. doi: 10.1182/bloodadvances.2022007263. PMID 35381071
- [Background] Hlavacek P, Guo JD, Rosenblatt L, Keshishian A, Russ C, Mardekian J, Ferri M, Poretta T, Yuce H, McBane R. Safety, effectiveness, and health care cost comparisons among elderly patients with venous thromboembolism prescribed warfarin or apixaban in the United States Medicare population. Curr Med Res Opin. 2019 Dec;35(12):2043-2051. doi: 10.1080/03007995.2019.1653067. Epub 2019 Sep 3. PMID 31387467
- [Background] Linkins LA, Choi PT, Douketis JD. Clinical impact of bleeding in patients taking oral anticoagulant therapy for venous thromboembolism: a meta-analysis. Ann Intern Med. 2003 Dec 2;139(11):893-900. doi: 10.7326/0003-4819-139-11-200312020-00007. PMID 14644891
- [Background] Aryal MR, Gosain R, Donato A, Yu H, Katel A, Bhandari Y, Dhital R, Kouides PA. Systematic review and meta-analysis of the efficacy and safety of apixaban compared to rivaroxaban in acute VTE in the real world. Blood Adv. 2019 Aug 13;3(15):2381-2387. doi: 10.1182/bloodadvances.2019000572. PMID 31405948
- [Background] Sindet-Pedersen C, Staerk L, Pallisgaard JL, Gerds TA, Berger JS, Torp-Pedersen C, Gislason GH, Olesen JB. Safety and effectiveness of rivaroxaban and apixaban in patients with venous thromboembolism: a nationwide study. Eur Heart J Cardiovasc Pharmacother. 2018 Oct 1;4(4):220-227. doi: 10.1093/ehjcvp/pvy021. PMID 29945162
- [Background] Catella J, Bertoletti L, Moustafa F, Nieto JA, Valle R, Pedrajas JM, Villalobos A, Quere I, Sarlon-Bartoli G, Monreal M; RIETE Investigators. Major gastrointestinal bleeding in patients receiving anticoagulant therapy for venous thromboembolism. Thromb Res. 2022 Jun;214:29-36. doi: 10.1016/j.thromres.2022.04.005. Epub 2022 Apr 13. PMID 35452869
- [Background] Dawwas GK, Leonard CE, Lewis JD, Cuker A. Risk for Recurrent Venous Thromboembolism and Bleeding With Apixaban Compared With Rivaroxaban: An Analysis of Real-World Data. Ann Intern Med. 2022 Jan;175(1):20-28. doi: 10.7326/M21-0717. Epub 2021 Dec 7. PMID 34871048
- [Background] Schulman S, Kakkar AK, Goldhaber SZ, Schellong S, Eriksson H, Mismetti P, Christiansen AV, Friedman J, Le Maulf F, Peter N, Kearon C; RE-COVER II Trial Investigators. Treatment of acute venous thromboembolism with dabigatran or warfarin and pooled analysis. Circulation. 2014 Feb 18;129(7):764-72. doi: 10.1161/CIRCULATIONAHA.113.004450. Epub 2013 Dec 16. PMID 24344086
- [Background] Schulman S, Kearon C, Kakkar AK, Schellong S, Eriksson H, Baanstra D, Kvamme AM, Friedman J, Mismetti P, Goldhaber SZ; RE-MEDY Trial Investigators; RE-SONATE Trial Investigators. Extended use of dabigatran, warfarin, or placebo in venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):709-18. doi: 10.1056/NEJMoa1113697. PMID 23425163
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Background] Prins MH, Lensing AW, Bauersachs R, van Bellen B, Bounameaux H, Brighton TA, Cohen AT, Davidson BL, Decousus H, Raskob GE, Berkowitz SD, Wells PS; EINSTEIN Investigators. Oral rivaroxaban versus standard therapy for the treatment of symptomatic venous thromboembolism: a pooled analysis of the EINSTEIN-DVT and PE randomized studies. Thromb J. 2013 Sep 20;11(1):21. doi: 10.1186/1477-9560-11-21. PMID 24053656
- [Background] Wells PS, Prins MH, Levitan B, Beyer-Westendorf J, Brighton TA, Bounameaux H, Cohen AT, Davidson BL, Prandoni P, Raskob GE, Yuan Z, Katz EG, Gebel M, Lensing AWA. Long-term Anticoagulation With Rivaroxaban for Preventing Recurrent VTE: A Benefit-Risk Analysis of EINSTEIN-Extension. Chest. 2016 Nov;150(5):1059-1068. doi: 10.1016/j.chest.2016.05.023. Epub 2016 Jun 1. PMID 27262225
- [Background] Agnelli G, Becattini C, Meyer G, Munoz A, Huisman MV, Connors JM, Cohen A, Bauersachs R, Brenner B, Torbicki A, Sueiro MR, Lambert C, Gussoni G, Campanini M, Fontanella A, Vescovo G, Verso M; Caravaggio Investigators. Apixaban for the Treatment of Venous Thromboembolism Associated with Cancer. N Engl J Med. 2020 Apr 23;382(17):1599-1607. doi: 10.1056/NEJMoa1915103. Epub 2020 Mar 29. PMID 32223112
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- [Background] Young AM, Marshall A, Thirlwall J, Chapman O, Lokare A, Hill C, Hale D, Dunn JA, Lyman GH, Hutchinson C, MacCallum P, Kakkar A, Hobbs FDR, Petrou S, Dale J, Poole CJ, Maraveyas A, Levine M. Comparison of an Oral Factor Xa Inhibitor With Low Molecular Weight Heparin in Patients With Cancer With Venous Thromboembolism: Results of a Randomized Trial (SELECT-D). J Clin Oncol. 2018 Jul 10;36(20):2017-2023. doi: 10.1200/JCO.2018.78.8034. Epub 2018 May 10. PMID 29746227
- [Background] Raskob G, Buller H, Prins M, Segers A, Shi M, Schwocho L, van Kranen R, Mercuri M; Hokusai-VTE Investigators. Edoxaban for the long-term treatment of venous thromboembolism: rationale and design of the Hokusai-venous thromboembolism study--methodological implications for clinical trials. J Thromb Haemost. 2013 Jul;11(7):1287-94. doi: 10.1111/jth.12230. PMID 23574579
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Raskob GE, van Es N, Verhamme P, Carrier M, Di Nisio M, Garcia D, Grosso MA, Kakkar AK, Kovacs MJ, Mercuri MF, Meyer G, Segers A, Shi M, Wang TF, Yeo E, Zhang G, Zwicker JI, Weitz JI, Buller HR; Hokusai VTE Cancer Investigators. Edoxaban for the Treatment of Cancer-Associated Venous Thromboembolism. N Engl J Med. 2018 Feb 15;378(7):615-624. doi: 10.1056/NEJMoa1711948. Epub 2017 Dec 12. PMID 29231094
- [Background] Douketis JD, Foster GA, Crowther MA, Prins MH, Ginsberg JS. Clinical risk factors and timing of recurrent venous thromboembolism during the initial 3 months of anticoagulant therapy. Arch Intern Med. 2000 Dec 11-25;160(22):3431-6. doi: 10.1001/archinte.160.22.3431. PMID 11112236
- [Background] Gitter MJ, Jaeger TM, Petterson TM, Gersh BJ, Silverstein MD. Bleeding and thromboembolism during anticoagulant therapy: a population-based study in Rochester, Minnesota. Mayo Clin Proc. 1995 Aug;70(8):725-33. doi: 10.4065/70.8.725. PMID 7630209
- [Background] Carrier M, Le Gal G, Wells PS, Rodger MA. Systematic review: case-fatality rates of recurrent venous thromboembolism and major bleeding events among patients treated for venous thromboembolism. Ann Intern Med. 2010 May 4;152(9):578-89. doi: 10.7326/0003-4819-152-9-201005040-00008. PMID 20439576
- [Background] Connolly SJ, Crowther M, Eikelboom JW, Gibson CM, Curnutte JT, Lawrence JH, Yue P, Bronson MD, Lu G, Conley PB, Verhamme P, Schmidt J, Middeldorp S, Cohen AT, Beyer-Westendorf J, Albaladejo P, Lopez-Sendon J, Demchuk AM, Pallin DJ, Concha M, Goodman S, Leeds J, Souza S, Siegal DM, Zotova E, Meeks B, Ahmad S, Nakamya J, Milling TJ Jr; ANNEXA-4 Investigators. Full Study Report of Andexanet Alfa for Bleeding Associated with Factor Xa Inhibitors. N Engl J Med. 2019 Apr 4;380(14):1326-1335. doi: 10.1056/NEJMoa1814051. Epub 2019 Feb 7. PMID 30730782
- [Background] Pollack CV Jr, Reilly PA, Weitz JI. Dabigatran Reversal with Idarucizumab. N Engl J Med. 2017 Oct 26;377(17):1691-2. doi: 10.1056/NEJMc1711337. No abstract available. PMID 29069562
- [Background] Held C, Hylek EM, Alexander JH, Hanna M, Lopes RD, Wojdyla DM, Thomas L, Al-Khalidi H, Alings M, Xavier D, Ansell J, Goto S, Ruzyllo W, Rosenqvist M, Verheugt FW, Zhu J, Granger CB, Wallentin L. Clinical outcomes and management associated with major bleeding in patients with atrial fibrillation treated with apixaban or warfarin: insights from the ARISTOTLE trial. Eur Heart J. 2015 May 21;36(20):1264-72. doi: 10.1093/eurheartj/ehu463. Epub 2014 Dec 12. PMID 25499871
- [Background] Klok FA, Niemann C, Dellas C, Hasenfuss G, Konstantinides S, Lankeit M. Performance of five different bleeding-prediction scores in patients with acute pulmonary embolism. J Thromb Thrombolysis. 2016 Feb;41(2):312-20. doi: 10.1007/s11239-015-1239-x. PMID 26091712
- [Background] Klok FA, Hosel V, Clemens A, Yollo WD, Tilke C, Schulman S, Lankeit M, Konstantinides SV. Prediction of bleeding events in patients with venous thromboembolism on stable anticoagulation treatment. Eur Respir J. 2016 Nov;48(5):1369-1376. doi: 10.1183/13993003.00280-2016. Epub 2016 Jul 28. PMID 27471209
- [Background] Thomopoulos KC, Mimidis KP, Theocharis GJ, Gatopoulou AG, Kartalis GN, Nikolopoulou VN. Acute upper gastrointestinal bleeding in patients on long-term oral anticoagulation therapy: endoscopic findings, clinical management and outcome. World J Gastroenterol. 2005 Mar 7;11(9):1365-8. doi: 10.3748/wjg.v11.i9.1365. PMID 15761977
- [Background] Morin J, Alayche M, Ghossein J, Delluc C, Siegal D, Wang TF, Delluc A. Source of upper gastrointestinal bleeding in cancer patients: A cross-sectional study. Thromb Res. 2022 Sep;217:9-11. doi: 10.1016/j.thromres.2022.06.009. Epub 2022 Jul 1. No abstract available. PMID 35810617
- [Background] Deitelzweig S, Keshishian A, Kang A, Dhamane AD, Luo X, Balachander N, Rosenblatt L, Mardekian J, Jiang J, Yuce H, Lip GYH. Burden of major gastrointestinal bleeding among oral anticoagulant-treated non-valvular atrial fibrillation patients. Therap Adv Gastroenterol. 2021 Mar 21;14:1756284821997352. doi: 10.1177/1756284821997352. eCollection 2021. PMID 33815568
- [Background] Sherwood MW, Nessel CC, Hellkamp AS, Mahaffey KW, Piccini JP, Suh EY, Becker RC, Singer DE, Halperin JL, Hankey GJ, Berkowitz SD, Fox KAA, Patel MR. Gastrointestinal Bleeding in Patients With Atrial Fibrillation Treated With Rivaroxaban or Warfarin: ROCKET AF Trial. J Am Coll Cardiol. 2015 Dec 1;66(21):2271-2281. doi: 10.1016/j.jacc.2015.09.024. PMID 26610874
- [Background] Candeloro M, van Es N, Cantor N, Schulman S, Carrier M, Ageno W, Aibar J, Donadini MP, Bavalia R, Arsenault MP, Coppens M, Ferrante N, D'Addezio A, Sormani S, Porreca E, Di Nisio M. Recurrent bleeding and thrombotic events after resumption of oral anticoagulants following gastrointestinal bleeding: Communication from the ISTH SSC Subcommittee on Control of Anticoagulation. J Thromb Haemost. 2021 Oct;19(10):2618-2628. doi: 10.1111/jth.15476. Epub 2021 Aug 8. PMID 34318606
- [Background] Ruff CT, Giugliano RP, Braunwald E, Hoffman EB, Deenadayalu N, Ezekowitz MD, Camm AJ, Weitz JI, Lewis BS, Parkhomenko A, Yamashita T, Antman EM. Comparison of the efficacy and safety of new oral anticoagulants with warfarin in patients with atrial fibrillation: a meta-analysis of randomised trials. Lancet. 2014 Mar 15;383(9921):955-62. doi: 10.1016/S0140-6736(13)62343-0. Epub 2013 Dec 4. PMID 24315724
- [Background] Schulman S, Gross PL, Ritchie B, Nahirniak S, Lin Y, Lieberman L, Carrier M, Crowther MA, Ghosh I, Lazo-Langner A, Zondag M; Study Investigators. Prothrombin Complex Concentrate for Major Bleeding on Factor Xa Inhibitors: A Prospective Cohort Study. Thromb Haemost. 2018 May;118(5):842-851. doi: 10.1055/s-0038-1636541. Epub 2018 Mar 21. PMID 29564837
- [Background] Majeed A, Agren A, Holmstrom M, Bruzelius M, Chaireti R, Odeberg J, Hempel EL, Magnusson M, Frisk T, Schulman S. Management of rivaroxaban- or apixaban-associated major bleeding with prothrombin complex concentrates: a cohort study. Blood. 2017 Oct 12;130(15):1706-1712. doi: 10.1182/blood-2017-05-782060. Epub 2017 Aug 23. PMID 28835439
- [Background] Gomez-Outes A, Alcubilla P, Calvo-Rojas G, Terleira-Fernandez AI, Suarez-Gea ML, Lecumberri R, Vargas-Castrillon E. Meta-Analysis of Reversal Agents for Severe Bleeding Associated With Direct Oral Anticoagulants. J Am Coll Cardiol. 2021 Jun 22;77(24):2987-3001. doi: 10.1016/j.jacc.2021.04.061. PMID 34140101
- [Background] Nieto JA, Solano R, Ruiz-Ribo MD, Ruiz-Gimenez N, Prandoni P, Kearon C, Monreal M; Riete Investigators. Fatal bleeding in patients receiving anticoagulant therapy for venous thromboembolism: findings from the RIETE registry. J Thromb Haemost. 2010 Jun;8(6):1216-22. doi: 10.1111/j.1538-7836.2010.03852.x. Epub 2010 Mar 12. PMID 20345727
- [Background] Little DHW, Sutradhar R, Cerasuolo JO, Perez R, Douketis J, Holbrook A, Paterson JM, Gomes T, Siegal DM. Rates of rebleeding, thrombosis and mortality associated with resumption of anticoagulant therapy after anticoagulant-related bleeding. CMAJ. 2021 Mar 1;193(9):E304-E309. doi: 10.1503/cmaj.201433. PMID 33649169
- [Background] Little D, Chai-Adisaksopha C, Hillis C, Witt DM, Monreal M, Crowther MA, Siegal DM. Resumption of anticoagulant therapy after anticoagulant-related gastrointestinal bleeding: A systematic review and meta-analysis. Thromb Res. 2019 Mar;175:102-109. doi: 10.1016/j.thromres.2019.01.020. Epub 2019 Jan 30. PMID 30743134
- [Background] Wang K, Li H, Kwong WJ, Antman EM, Ruff CT, Giugliano RP, Cohen DJ, Magnuson EA; ENGAGE AF-TIMI 48 Trial Investigators. Impact of Spontaneous Extracranial Bleeding Events on Health State Utility in Patients with Atrial Fibrillation: Results from the ENGAGE AF-TIMI 48 Trial. J Am Heart Assoc. 2017 Aug 11;6(8):e006703. doi: 10.1161/JAHA.117.006703. PMID 28862934
- [Background] Targownik LE, Fisher DA, Saini SD. AGA Clinical Practice Update on De-Prescribing of Proton Pump Inhibitors: Expert Review. Gastroenterology. 2022 Apr;162(4):1334-1342. doi: 10.1053/j.gastro.2021.12.247. Epub 2022 Feb 17. PMID 35183361
- [Background] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Background] Moayyedi P, Eikelboom JW, Bosch J, Connolly SJ, Dyal L, Shestakovska O, Leong D, Anand SS, Stork S, Branch KRH, Bhatt DL, Verhamme PB, O'Donnell M, Maggioni AP, Lonn EM, Piegas LS, Ertl G, Keltai M, Cook Bruns N, Muehlhofer E, Dagenais GR, Kim JH, Hori M, Steg PG, Hart RG, Diaz R, Alings M, Widimsky P, Avezum A, Probstfield J, Zhu J, Liang Y, Lopez-Jaramillo P, Kakkar A, Parkhomenko AN, Ryden L, Pogosova N, Dans A, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik T, Vinereanu D, Tonkin AM, Lewis BS, Felix C, Yusoff K, Metsarinne K, Fox KAA, Yusuf S; COMPASS Investigators. Pantoprazole to Prevent Gastroduodenal Events in Patients Receiving Rivaroxaban and/or Aspirin in a Randomized, Double-Blind, Placebo-Controlled Trial. Gastroenterology. 2019 Aug;157(2):403-412.e5. doi: 10.1053/j.gastro.2019.04.041. Epub 2019 May 2. PMID 31054846
- [Background] Dong Y, He S, Li X, Zhou Z. Prevention of nNon-Vitamin K Oral Anticoagulants-Related Gastrointestinal Bleeding With Acid Suppressants: A Systematic Review and Meta-Analysis. Clin Appl Thromb Hemost. 2022 Jan-Dec;28:10760296211064897. doi: 10.1177/10760296211064897. PMID 35037779
- [Background] Bang CS, Joo MK, Kim BW, Kim JS, Park CH, Ahn JY, Lee JH, Lee BE, Yang HJ, Cho YK, Park JM, Kim BJ, Jung HK; Korean College of Helicobacter and Upper Gastrointestinal Research. The Role of Acid Suppressants in the Prevention of Anticoagulant-Related Gastrointestinal Bleeding: A Systematic Review and Meta-Analysis. Gut Liver. 2020 Jan 15;14(1):57-66. doi: 10.5009/gnl19009. PMID 30974930
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Kaatz S, Ahmad D, Spyropoulos AC, Schulman S; Subcommittee on Control of Anticoagulation. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Nov;13(11):2119-26. doi: 10.1111/jth.13140. No abstract available. PMID 26764429
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Spence J, Bosch J, Chongsi E, Lee SF, Thabane L, Mendoza P, Belley-Cote E, Whitlock R, Brady K, McIntyre WF, Lamy A, Devereaux PJ. Standardized Assessment of Global activities in the Elderly scale in adult cardiac surgery patients. Br J Anaesth. 2021 Oct;127(4):539-546. doi: 10.1016/j.bja.2021.05.037. Epub 2021 Jul 28. PMID 34330417
- [Background] Forbes N, Elmunzer BJ, Keswani RN, Hilsden RJ, Hall M, Anderson JT, Arvanitakis M, Chen YI, Duloy A, Elta GH, Maranki JL, Mergener K, Petersen BT, Sethi A, Siersema PD, Smith ZL, Telford JJ, Tse F, Cotton PB, Wani S. Consensus-based development of a causal attribution system for post-ERCP adverse events. Gut. 2022 Jul 11:gutjnl-2022-328059. doi: 10.1136/gutjnl-2022-328059. Online ahead of print. No abstract available. PMID 35817552
- [Background] Hilsden RJ, Maxwell CM, Forbes N, Bridges RJ, Rostom A, Dube C, Boyne D, Brenner D, Heitman SJ. Development of a definition and rules for causal attribution of post-colonoscopy bleeding. PLoS One. 2020 Jul 23;15(7):e0235902. doi: 10.1371/journal.pone.0235902. eCollection 2020. PMID 32701949
- [Background] Le Gal G, Carrier M, Castellucci LA, Cuker A, Hansen JB, Klok FA, Langlois NJ, Levy JH, Middeldorp S, Righini M, Walters S; ISTH CDE Task Force. Development and implementation of common data elements for venous thromboembolism research: on behalf of SSC Subcommittee on official Communication from the SSC of the ISTH. J Thromb Haemost. 2021 Jan;19(1):297-303. doi: 10.1111/jth.15138. PMID 33405381